CLINICAL TRIAL: NCT00625911
Title: Ketamine Improves Post-Thoracotomy Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Avi A Weinbroum, MD, Tel Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASMC-01-AW-114-CTIL
Record Dates: First submitted 2008-02-08; First posted 2008-02-29 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2008-02

CONDITIONS: Post Operative Pain
Keywords: thoracotomy; minimally invasive direct coronary artery bypass; ketamine; pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Morphine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- morphine only (Active Comparator): standard analgesia protocol
  Interventions: Drug: morphine
- morphine ketamine (Experimental): alterantive regimen for intravenous patient controlled analgesia
  Interventions: Drug: morphine ketamine

INTERVENTIONS:
Drug: morphine — intravenous patient controlled analgesia, standard protocol
  Arms: morphine only
Drug: morphine ketamine — low dose ketamine added to 2/3 standard dose of morphine
  Other Names: ketalar
  Arms: morphine ketamine

SUMMARY:
Thoracotomy for lung tumor or for minimally invasive direct coronary artery bypass (MIDCAB) surgery, may be associated with debilitating pain. Ketamine was shown to enhance opioid antinociception and prevent opioid resistance. We hypothesize that ketamine given with morphine would lower morphine consumption and narcotic related side effects after thoracotomy and provide superior analgesia to morphine given alone.

DETAILED DESCRIPTION:
We planned a prospective, randomomized, double blind study of 2 pain management protocols in consecutive patients undergoing thoracotomy for MIDCAB or lung tumor resection over a 6 month period. After patients emerged from a standardized general anesthetic and when objectively awake and complaining of pain >5/10 on a visual analogue pain scale, they were connected to an intravenous patient controlled analgesia regimen. The regimen was assigned randomly to be either morphine alone (1.5 mg per dose, lockout interval of 7 minutes) or morphine plus ketamine (1.0 mg morphine plus 5 mg ketamine per dose, same lockout interval). Rescue diclofenac was available to both groups. Follow-up lasted 4 hours.

We planned to monitor and compare pain scores, wakefulness scores, hemodynamic and respiratory parameters as well as total morphine consumption and incidence of side effects and complications. All monitoring and recording was done by blinded nurses and intensive care physicians.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients scheduled for elective minimally invasive direct coronary artery bypass (MIDCAB) or for lung resection via anterolateral thoracotomy during a 6-month period (Sep 2001-March 2002)

Exclusion Criteria:

Exclusion criteria were:

* American Society of Anesthesiologists (ASA) physical class ≥3, Emergency operations,
* Q-wave myocardial infarct occurring during the previous 3 weeks, or poor left ventricular function (e.g., ejection fraction [EF] <30% by echocardiography or angiography).

Other exclusion criteria were:

* A body mass index >35 kg/m2,
* Past or current neuropathy or psychological disturbances,
* The use of centrally active drugs,
* Chronic liver or renal failure requiring dialysis,
* A FEV1/FVC <70%,
* Allergy to ketamine, morphine or non steroidal anti inflammatory drugs (NSAIDs),
* Clotting abnormalities,
* A platelets count <70000/mm3,
* A white blood count <3000>14000/mm3,
* Uncontrolled diabetes mellitus or fasting blood glucose >250 g/dl,
* Evidence of sepsis or infection up to one week prior to randomization.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2001-09; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
pain score | 4 hours

SECONDARY OUTCOMES:
hemodynamic and respiratory parameters, side effects | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Avi A Weinbroum, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Nesher N, Ekstein MP, Paz Y, Marouani N, Chazan S, Weinbroum AA. Morphine with adjuvant ketamine vs higher dose of morphine alone for immediate postthoracotomy analgesia. Chest. 2009 Jul;136(1):245-252. doi: 10.1378/chest.08-0246. Epub 2008 Aug 27. PMID 18753471